CLINICAL TRIAL: NCT00852826
Title: Value of a Hemostatic and Sealing Agent for Preventing Seroma After Axillary Lymphadenectomy
Brief Title: Evaluation of a Hemostatic and Sealing Agent to Prevent Surgical Complications After Axillary Lymphadenectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LFN001/08
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Seroma
Keywords: axillary seroma; axillary lymphadenectomy; morbidity; morbidity postlymphadenectomy; Lymphadenectomy
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Sham Comparator): Standard axillary lymphadenectomy
  Interventions: Procedure: Standard axillary lymphadenectomy
- 2 (Experimental): Three patches of collagen sponge coated with human coagulation factors (TachoSil®, Nycomed Pharma, AS) were perpendicularly placed at the end of lymphadenectomy on the axillary neurovascular bundle, thoracodorsal pedicle, and costal wall, covering the axillary walls
  Interventions: Procedure: Collagen sponge coated with human coagulation factors

INTERVENTIONS:
Procedure: Standard axillary lymphadenectomy — Standard axillary lymphadenectomy
  Arms: 1
Procedure: Collagen sponge coated with human coagulation factors — Three patches of collagen sponge coated with human coagulation factors (TachoSil®, Nycomed Pharma, AS) were perpendicularly placed at the end of lymphadenectomy on the axillary neurovascular bundle, thoracodorsal pedicle, and costal wall, covering the axillary walls
  Other Names: TachoSil(R), Nycomed Pharma, AS.
  Arms: 2

SUMMARY:
This study was intended to assess the value of a hemostatic and sealing agent, a collagen sponge coated with human coagulation factors (fibrinogen and thrombin) (TachoSil®), for decreasing occurrence of seroma after axillary lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with axillary lymphadenectomies performed for oncological conditions.

Exclusion Criteria:

* Patients that did not want to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01; Study Completion 2008-11

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Piñero, MD PhD, Principal Investigator
Locations (1):
- Hospital Universitario "Virgen de la Arrixaca", Murcia, Murcia, Spain